CLINICAL TRIAL: NCT01275885
Title: Vitamin D Intervention in Infants - Pilot
Acronym: VIDI-P
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Sture Andersson, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: T1040D0038; 2009-015940-40 (EudraCT Number)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Vitamin D; Supplementation
Keywords: cholecalciferol; infant; bone mineral density
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Vitamin D3 10µg (Active Comparator)
  Interventions: Dietary Supplement: cholecalciferol (D3)
- Vitamin D3 30µg (Active Comparator)
  Interventions: Dietary Supplement: cholecalciferol (D3)
- Vitamin D3 40µg (Active Comparator)
  Interventions: Dietary Supplement: cholecalciferol (D3)

INTERVENTIONS:
Dietary Supplement: cholecalciferol (D3) — 10µg (400 IU) orally daily for 10 weeks
  Arms: Vitamin D3 10µg
Dietary Supplement: cholecalciferol (D3) — 30µg (1200 IU) orally daily for 10 weeks
  Arms: Vitamin D3 30µg
Dietary Supplement: cholecalciferol (D3) — 40µg (1600 IU) orally daily for 10 weeks
  Arms: Vitamin D3 40µg

SUMMARY:
The aims of the present study are to evaluate the concentrations of vitamin D in the plasma and of calcium in the plasma and in the urine as well as to evaluate bone mineral density using peripheral quantitative computed tomography (pQCT), after supplementation of vitamin D with 30µg (1200 IU) and 40µg (1600 IU), in comparison with currently recommended supplementation of vitamin D with 10µg (400 IU). In this pilot study supplementation is given to infants from 2 weeks of age to 3 months of age.

DETAILED DESCRIPTION:
Vitamin D deficiency is common around the world. In Finland vitamin D levels are low in all age groups. Especially infants are predisposed to vitamin D deficiency. Partly this is due to low exposure to sunlight but mainly it is due to low dietary intake of vitamin D. Vitamin D prophylaxis was introduced in Finland in the 1950´s to overcome rickets. However, the recommended dose has decreased from 50µg (2000 IU) in the 1960´s to 10µg (400 IU) from beginning of the 1990´s. The serum concentration of 25-hydroxyvitamin D (S-25OHD) is used as a marker of vitamin D status in the body. Although there is no consensus of optimal concentration of S-25OHD, it has been proposed that concentrations lower than 50 nmol/l indicate deficiency. According to recent findings on 25-OHD concentrations in Finnish children, currently recommended intake of vitamin D is inadequate.

ELIGIBILITY:
Inclusion Criteria:

* healthy Caucasian women with an uneventful pregnancy
* healthy infants born at term and appropriate for gestational age

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
S-25OHD concentration after vitamin D supplementation to infants | after 10 weeks of supplementation
  The primary endpoint is the concentration of 25OHD in serum after daily supplementation with vitamin D (10µg / 30µg / 40µg orally). Vitamin D supplementation is given to infants from 2 weeks of age to 3 months of age.

SECONDARY OUTCOMES:
concentration of calcium in the plasma and in the urine | after 10 weeks of supplementation
  Incidence of hypercalcemia and hypercalciuria in infants after daily supplementation with vitamin D (10µg / 30µg / 40µg orally).
bone mineral density | after 10 weeks of supplementation
  Measurement of bone mineral density using peripheral quantitative computed tomography (pQCT), after daily supplementation with vitamin D (10µg / 30µg / 40µg orally).

CONTACTS AND LOCATIONS:
Overall Officials: Sture Andersson, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Hospital for Children and Adolescents, Helsinki University Central Hospital, Helsinki, Finland